CLINICAL TRIAL: NCT03984149
Title: Prevalence and Mutation Rate of Lipa Gene in LIPIGEN Subjects With Clinical Diagnosis of FH
Brief Title: Lipa Gene Mutation in PED-LIPIGEN (Pediatric FH Subjects)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione SISA (Societa Italiana per lo Studio della Arteriosclerosi) (Other)
Responsible Party: Sponsor
Other Study IDs: LIPIGEN-002
Record Dates: First submitted 2019-05-21; First posted 2019-06-12 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Lysosomal Acid Lipase Deficiency
Keywords: Atherosclerosis; Familial hypercholesterolemia; LIPA; Lysosomal acid lipase deficiency; Wolman disease
MeSH Terms: conditions — Wolman Disease; Atherosclerosis; Hyperlipoproteinemia Type II | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Venous blood samples were taken after 12 hours of fasting. Serum total cholesterol, triglycerides and HDL-cholesterol levels were measured in a centralized laboratory using enzymatic methods.
  DNA samples, serum, plasma and whole blood were aliquoted and preserved at -80°C.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FH pediatric patients: 1000 clinically diagnosed FH pediatric patients (age <18 years) included in the LIPIGEN (Lipid TransPort Disorders italian Genetic Network) database
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — Observational study: There is no intervention.

SUMMARY:
Familial Hypercholesterolemia (FH) is a monogenic autosomal dominant disease also known as Autosomal Dominant Hypercholesterolemia - ADH) that leads to dramatically increased levels of Low Density Lipoprotein (LDL) and total cholesterol associated to tendon xanthomas, xanthelasma, corneal arcus, premature atherosclerosis and to an increased risk of coronary artery disease (CAD) and myocardial infarction.

FH is mainly caused by mutations in genes encoding for proteins affecting hepatic LDL cholesterol uptake including the LDL receptor (LDLR) gene or the gene encoding the only apolipoprotein of LDL, the apolipoprotein B (APOB), or the gene encoding a protease regulating LDLR levels on the cell membrane Lysosomal Acid Lipase A (LIPA) gene encode for Lysosomal acid lipase (LAL) enzyme responsible for hydrolyzing cholesterol esters and triglycerides that are delivered to lysosomes. Mutations in LIPA that completely inactivate LAL are the molecular cause of Wolman disease, a rapidly lethal disease of infancy while mutations in LIPA that result in residual enzymatic activity of LAL are responsible of a disorder characterized by a less severe phenotype known as cholesterol ester storage disease (CESD). Patients with CESD usually show a phenotype characterized by hepatic disease and mixed hyperlipidemia with elevated levels of LDL-C and triglycerides (TG) and decreased HDL-C levels.

A broader phenotypic presentation for loss of function mutations in LIPA suggests that LIPA mutations may be considered in patients with apparently monogenic FH in whom mutations in the known candidate genes are not detectable.

The project is aimed to evaluate the prevalence and the mutation rate of LIPA gene in subjects with a clinical diagnosis of FH and already genetically characterized in whom pathogenic mutations in the known candidate genes have not been identified. The analysis will be performed in about 250 FH pediatric subjects and putative causal mutations will be also tested for co-segregation in available families in affected and unaffected members.

DETAILED DESCRIPTION:
Lysosomal acid lipase (LAL) is encoded by LIPA gene located on chromosome 10q23.3-q23 and consists of 10 exons. LIPA mRNA (messenger RiboNucleic Acid) (GenBank accession number NM_000235) is 2782 bp long and encodes a mature protein of 375 residues (GenBank accession number NP_000226). The sequencing of all 10 exons of LIPA gene will consist of 10 PCR (Polymerase Chain Reaction) amplification reactions (for the 10 exons and the proximal promoter) followed by 20 sequence reactions (forward and reverse sequencing) with appropriate primers designed to include the intron-exon boundaries. This analysis will be performed in about 250 FH pediatric subjects as specified in project description.

The sequencing work will be performed taking advantage of 2 automated 8 capillaries automated DNA Sequencer (3500 Genetic Analyzer, Thermo Fisher Scientific, Monza, Italy) currently available in the laboratory of the Units involved in the project.

In case of identification of unreported sequence variants, the presence of these mutations will be assessed in a sample of at least 100 normolipidemic subjects of the population, in order to define whether the nucleotide changes are rare sequence variations (with a putative functional effect) or represent common polymorphisms. In case of finding of rare variants in the coding regions, an in silico analysis will be performed by using two different softwares (Polyphen, http://genetics.bwh.harvard.edu/pph/ and Panther, http://www.pantherdb.org/) to predict the putative damaging role of the mutations on the protein. In case of intronic variants, the specifically designed software Automated Splice Site Analysis will be applied (https://www.splice.uwo.ca/).

Putative causal mutations will be also tested for co-segregation in available families in affected and unaffected members.

In order to test the effect of variants on enzyme activity LAL-activity will be assayed with dried blood spot (DBS) technique using the inhibitors Lalistat 2 in carriers and non carriers of these mutations belonging to available kindred.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric subjects (<18 years old) with a clinical diagnosis of FH and without identified pathogenic mutations in the known candidate genes.

Exclusion Criteria:

* Subjects with a clinical diagnosis of FH with identified pathogenic mutations in the known candidate genes.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Clinically diagnosed FH pediatric patients (age <18 years) included in the Lipid TransPort Disorders italian Genetic Network (LIPIGEN) database, already genetically characterized.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of patients with mutations of LIPA gene among clinically diagnosed FH subjects | 2 years from start of the study
  Percentage of patients with at least one mutation of LIPA gene among clinically diagnosed FH subjects according to a "Dutch Lipid Clinic Network" score of 6 or above

SECONDARY OUTCOMES:
Frequency of specific mutations of LIPA gene among clinically diagnosed FH subjects | 2 years from start of the study
  Numbers of patients carrying specific mutations of LIPA gene among clinically diagnosed FH subjects for each mutation identified by sequencing of all 10 exons of LIPA gene.

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Averna, Study Director — Fondazione SISA
Locations (4):
- Italy (4):
  - CENTRO PER LO STUDIO DELL'ATEROSCLEROSI - Ospedale Bassini, Cinisello Balsamo, Mi
  - Laboratorio di biochimica delle lipoproteine - DIPARTIMENTO DI SCIENZE BIOMEDICHE, Modena
  - Centro Di Riferimento Regionale Per La Prevenzione, Diagnosi E Cura Delle Malattie Rare Del Metabolismo, Palermo
  - Centro Per L'Arteriosclerosi Dipartimento Di Medicina Interna E Specialità Mediche, Roma

IPD SHARING:
Plan to Share IPD: Yes
Upon preventive request for a scientific collaboration
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: For three years from the end of the study
Access Criteria: Upon preventive request for a scientific collaboration

REFERENCES:
- [Background] ABRAMOV A, SCHORR S, WOLMAN M. Generalized xanthomatosis with calcified adrenals. AMA J Dis Child. 1956 Mar;91(3):282-6. doi: 10.1001/archpedi.1956.02060020284010. No abstract available. PMID 13301142
- [Background] Bernstein DL, Hulkova H, Bialer MG, Desnick RJ. Cholesteryl ester storage disease: review of the findings in 135 reported patients with an underdiagnosed disease. J Hepatol. 2013 Jun;58(6):1230-43. doi: 10.1016/j.jhep.2013.02.014. Epub 2013 Feb 26. PMID 23485521
- [Background] Bertolini S, Pisciotta L, Rabacchi C, Cefalu AB, Noto D, Fasano T, Signori A, Fresa R, Averna M, Calandra S. Spectrum of mutations and phenotypic expression in patients with autosomal dominant hypercholesterolemia identified in Italy. Atherosclerosis. 2013 Apr;227(2):342-8. doi: 10.1016/j.atherosclerosis.2013.01.007. Epub 2013 Jan 19. PMID 23375686
- [Background] Burke JA, Schubert WK. Deficient activity of hepatic acid lipase in cholesterol ester storage disease. Science. 1972 Apr 21;176(4032):309-10. doi: 10.1126/science.176.4032.309. PMID 5019788
- [Background] Futema M, Plagnol V, Li K, Whittall RA, Neil HA, Seed M; Simon Broome Consortium; Bertolini S, Calandra S, Descamps OS, Graham CA, Hegele RA, Karpe F, Durst R, Leitersdorf E, Lench N, Nair DR, Soran H, Van Bockxmeer FM; UK10K Consortium; Humphries SE. Whole exome sequencing of familial hypercholesterolaemia patients negative for LDLR/APOB/PCSK9 mutations. J Med Genet. 2014 Aug;51(8):537-44. doi: 10.1136/jmedgenet-2014-102405. Epub 2014 Jul 1. PMID 24987033
- [Background] Hamilton J, Jones I, Srivastava R, Galloway P. A new method for the measurement of lysosomal acid lipase in dried blood spots using the inhibitor Lalistat 2. Clin Chim Acta. 2012 Aug 16;413(15-16):1207-10. doi: 10.1016/j.cca.2012.03.019. Epub 2012 Mar 29. PMID 22483793
- [Background] Hopkins PN, Toth PP, Ballantyne CM, Rader DJ; National Lipid Association Expert Panel on Familial Hypercholesterolemia. Familial hypercholesterolemias: prevalence, genetics, diagnosis and screening recommendations from the National Lipid Association Expert Panel on Familial Hypercholesterolemia. J Clin Lipidol. 2011 Jun;5(3 Suppl):S9-17. doi: 10.1016/j.jacl.2011.03.452. Epub 2011 Apr 3. No abstract available. PMID 21600530
- [Background] Nordestgaard BG, Chapman MJ, Humphries SE, Ginsberg HN, Masana L, Descamps OS, Wiklund O, Hegele RA, Raal FJ, Defesche JC, Wiegman A, Santos RD, Watts GF, Parhofer KG, Hovingh GK, Kovanen PT, Boileau C, Averna M, Boren J, Bruckert E, Catapano AL, Kuivenhoven JA, Pajukanta P, Ray K, Stalenhoef AF, Stroes E, Taskinen MR, Tybjaerg-Hansen A; European Atherosclerosis Society Consensus Panel. Familial hypercholesterolaemia is underdiagnosed and undertreated in the general population: guidance for clinicians to prevent coronary heart disease: consensus statement of the European Atherosclerosis Society. Eur Heart J. 2013 Dec;34(45):3478-90a. doi: 10.1093/eurheartj/eht273. Epub 2013 Aug 15. PMID 23956253
- [Background] Patrick AD, Lake BD. Deficiency of an acid lipase in Wolman's disease. Nature. 1969 Jun 14;222(5198):1067-8. doi: 10.1038/2221067a0. No abstract available. PMID 5787090
- [Background] Risk of fatal coronary heart disease in familial hypercholesterolaemia. Scientific Steering Committee on behalf of the Simon Broome Register Group. BMJ. 1991 Oct 12;303(6807):893-6. doi: 10.1136/bmj.303.6807.893. PMID 1933004
- [Background] Stitziel NO, Fouchier SW, Sjouke B, Peloso GM, Moscoso AM, Auer PL, Goel A, Gigante B, Barnes TA, Melander O, Orho-Melander M, Duga S, Sivapalaratnam S, Nikpay M, Martinelli N, Girelli D, Jackson RD, Kooperberg C, Lange LA, Ardissino D, McPherson R, Farrall M, Watkins H, Reilly MP, Rader DJ, de Faire U, Schunkert H, Erdmann J, Samani NJ, Charnas L, Altshuler D, Gabriel S, Kastelein JJ, Defesche JC, Nederveen AJ, Kathiresan S, Hovingh GK; National Heart, Lung, and Blood Institute GO Exome Sequencing Project. Exome sequencing and directed clinical phenotyping diagnose cholesterol ester storage disease presenting as autosomal recessive hypercholesterolemia. Arterioscler Thromb Vasc Biol. 2013 Dec;33(12):2909-14. doi: 10.1161/ATVBAHA.113.302426. Epub 2013 Sep 26. PMID 24072694
- [Background] Talmud PJ, Futema M, Humphries SE. The genetic architecture of the familial hyperlipidaemia syndromes: rare mutations and common variants in multiple genes. Curr Opin Lipidol. 2014 Aug;25(4):274-81. doi: 10.1097/MOL.0000000000000090. PMID 24977977
- [Background] Williams RR, Hunt SC, Schumacher MC, Hegele RA, Leppert MF, Ludwig EH, Hopkins PN. Diagnosing heterozygous familial hypercholesterolemia using new practical criteria validated by molecular genetics. Am J Cardiol. 1993 Jul 15;72(2):171-6. doi: 10.1016/0002-9149(93)90155-6. PMID 8328379
- See also: Familial hypercholesterolaemia (FH) : report of a second World Health Organization (WHO) consultation, Geneva, 4 September 1998 — https://apps.who.int/iris/handle/10665/66346